CLINICAL TRIAL: NCT04592913
Title: A Randomized, Double-blind, Placebo-controlled, Phase III Study of Neoadjuvant-Adjuvant Durvalumab and FLOT Chemotherapy Followed by Adjuvant Durvalumab in Patients With Resectable Gastric and Gastroesophageal Junction Cancer (GC/GEJC)
Brief Title: Assessing Durvalumab and FLOT Chemotherapy in Resectable Gastric and Gastroesophageal Junction Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D910GC00001; 2019-001555-40 (EudraCT Number)
Record Dates: First submitted 2020-08-26; First posted 2020-10-19 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Gastrointestinal Neoplasms; Esophagogastric Junction
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — durvalumab

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind, Placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm B (Placebo Comparator): placebo product and FLOT chemotherapy
  Interventions: Drug: FLOT chemotherapy
- Arm A (Experimental): Durvalumab and FLOT chemotherapy
  Interventions: Drug: Durvalumab; Drug: FLOT chemotherapy

INTERVENTIONS:
Drug: Durvalumab — Human monoclonal antibody
  Arms: Arm A
Drug: FLOT chemotherapy — A combination treatment made up of flurouroacil + leucovorin + oxaliplatin + docetaxel

SUMMARY:
This is a Global Study of Neoadjuvant-Adjuvant Durvalumab or Placebo and FLOT Chemotherapy Followed by Adjuvant Durvalumab or Placebo in Patients with Resectable Gastric and Gastroesophageal Cancer (GC/GEJC) (MATTERHORN).

DETAILED DESCRIPTION:
This study investigates treatment of durvalumab or placebo therapy combined with FLOT chemotherapy (flurouroacil + leucovorin + oxaliplatin + docetaxel) given before surgery (neoadjuvant) and durvalumab or placebo therapy combined with FLOT chemotherapy after surgery (adjuvant), will work and be safe for the treatment of resectable (removable by surgery) gastric or gastroesophageal cancer, and also to better understand the studied disease and associated health problems.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients with histologically documented gastric or gastroesophageal junction adenocarcinoma with resectable disease (Stage II or higher per AJCC 8th edition).
* Patients must undergo radical surgery.
* No prior anti-cancer therapy for the current malignancy.
* World Health Organization (WHO)/ECOG performance status of 0 or 1 at enrollment.
* Adequate organ and marrow function.
* Availability of tumor sample prior to study entry.
* Must have a life expectancy of at least 24 weeks.

Key Exclusion Criteria:

* Patients with peritoneal dissemination or distant metastasis.
* Patients with adenosquamous cell carcinoma, squamous cell carcinoma, or GI stromal tumor.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab.
* Contra-indication to any of the study drugs.
* History of allogeneic organ transplantation.

Ages: 18 Years to 200 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 957 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2027-09-27 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | Up to 5 years
  EFS is the time from date of randomization until the date of disease progression or death.

SECONDARY OUTCOMES:
To compare Arm A relative to Arm B on overall survival (OS) | Up to 5 years
  Overall survival is length of time from randomization until the date of death due to any cause.
To compare Arm A relative to Arm B on pathological complete response (pCR) rate | Up to 5 years
  pCR rate is the proportion of patients who have no residual viable tumor in the resected specimens.

CONTACTS AND LOCATIONS:
Locations (132):
- United States (15):
  - Research Site, Duarte, California
  - Research Site, Los Angeles, California
  - Research Site, Sylmar, California
  - Research Site, St. Petersburg, Florida
  - Research Site, Tallahassee, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Fort Wayne, Indiana
  - Research Site, Louisville, Kentucky
  - Research Site, Boston, Massachusetts
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Lancaster, Texas
  - Research Site, Seattle, Washington
- Argentina (4):
  - Research Site, Buenos Aires
  - Research Site, Ciudad Autonoma Buenos Aires
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Rosario
- Belgium (5):
  - Research Site, Charleroi
  - Research Site, Edegem
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Roeselare
- Brazil (6):
  - Research Site, Barretos
  - Research Site, Natal
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Canada (6):
  - Research Site, Edmonton, Alberta
  - Research Site, North York, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Montreal
- Chile (4):
  - Research Site, La Serena
  - Research Site, Santiago
  - Research Site, Talca
  - Research Site, Temuco
- Denmark (3):
  - Research Site, Aalborg
  - Research Site, København Ø
  - Research Site, Odense
- France (10):
  - Research Site, Avignon
  - Research Site, Besançon
  - Research Site, Brest
  - Research Site, Dijon
  - Research Site, Lyon
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Rennes
- Germany (11):
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Frankfurt
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Heilbronn
  - Research Site, Jena
  - Research Site, Mainz Am Rhein
  - Research Site, München
  - Research Site, Schweinfurt
  - Research Site, Tübingen
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Győr
  - Research Site, Kecskemét
  - Research Site, Szekszárd
  - Research Site, Szolnok
- Japan (18):
  - Research Site, Chūōku
  - Research Site, Hidaka-shi
  - Research Site, Hirakata-shi
  - Research Site, Hiroshima
  - Research Site, Kashiwa
  - Research Site, Kitaadachi-gun
  - Research Site, Kochi
  - Research Site, Kurume-shi
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Ogaki-shi
  - Research Site, Osaka
  - Research Site, Suita-shi
  - Research Site, Sunto-gun
  - Research Site, Tokyo
  - Research Site, Toyoake-shi
  - Research Site, Wakayama
  - Research Site, Yokohama
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Eindhoven
  - Research Site, Rotterdam
- Peru (3):
  - Research Site, Bellavista
  - Research Site, Lima
  - Research Site, San Isidro
- Poland (6):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Poznan
  - Research Site, Warsaw
- Russia (5):
  - Research Site, Kaluga
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Obninsk
  - Research Site, Saint Petersburg
- South Korea (3):
  - Research Site, Hwasun-gun
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (7):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Ourense
  - Research Site, Santander
  - Research Site, Seville
  - Research Site, Valencia
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan
- Turkey (Türkiye) (5):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Erzurum
  - Research Site, Istanbul
  - Research Site, Samsun
- United Kingdom (8):
  - Research Site, Cambridge
  - Research Site, Dundee
  - Research Site, Glasgow
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Oxford
  - Research Site, Surrey

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Janjigian YY, Al-Batran SE, Wainberg ZA, Muro K, Molena D, Van Cutsem E, Hyung WJ, Wyrwicz L, Oh DY, Omori T, Moehler M, Garrido M, Oliveira SCS, Liberman M, Oliden VC, Smyth EC, Stein A, Bilici M, Alvarenga ML, Kozlov V, Rivera F, Kawazoe A, Serrano O, Heilbron E, Negro A, Kurland JF, Tabernero J; MATTERHORN Investigators. Perioperative Durvalumab in Gastric and Gastroesophageal Junction Cancer. N Engl J Med. 2025 Jul 17;393(3):217-230. doi: 10.1056/NEJMoa2503701. Epub 2025 Jun 1. PMID 40454643
- [Derived] Chang X, Ge X, Zhang Y, Xue X. The current management and biomarkers of immunotherapy in advanced gastric cancer. Medicine (Baltimore). 2022 May 27;101(21):e29304. doi: 10.1097/MD.0000000000029304. PMID 35623069
- [Derived] Janjigian YY, Van Cutsem E, Muro K, Wainberg Z, Al-Batran SE, Hyung WJ, Molena D, Marcovitz M, Ruscica D, Robbins SH, Negro A, Tabernero J. MATTERHORN: phase III study of durvalumab plus FLOT chemotherapy in resectable gastric/gastroesophageal junction cancer. Future Oncol. 2022 Jun;18(20):2465-2473. doi: 10.2217/fon-2022-0093. Epub 2022 May 10. PMID 35535555
- [Derived] Cowzer D, Janjigian YY. Top advances in esophageal/gastroesophageal junction cancers in 2021. Cancer. 2022 May 15;128(10):1894-1899. doi: 10.1002/cncr.34140. Epub 2022 Feb 18. No abstract available. PMID 35179774